CLINICAL TRIAL: NCT05558774
Title: Long-term Echocardiographic and Clinical Outcomes After Percutaneous Closure of Patent Foramen Ovale
Brief Title: Long-term Outcomes After Percutaneous Closure of PFO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MC Medicor (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Medicor-PFO
Record Dates: First submitted 2022-09-04; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Foramen Ovale, Patent; Echocardiography; Embolic Stroke; Atrial Fibrillation
Keywords: patent foramen ovale; transthoracic echocardiography; cerebrovascular insult; transient ischemic attack; atrial fibrillation
MeSH Terms: conditions — Foramen Ovale, Patent; Embolic Stroke; Atrial Fibrillation; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
International medical centre Medicor from Slovenia has reported 306 successful percutaneous closures of patent foramen ovale (PFO) from October 2006 till June 2022. The investigators are going to follow-up the participants clinically and with contrast transthoracic echocardiography (TTE) to define the percentage of functional percutaneous closure. The latter is defined with the number (ten or less) of contrast-bubbles in the left atrium during Valsalva maneuver and contrast (agitated saline) application. The clinical follow-up will show the recurrence of embolic events (cerebrovascular insults, transient ischemic attacks) after percutaneous closure. In addition all of the participants are going to be screened for atrial fibrillation. The patients with moderate residual shunts (more than ten bubbles in the left atrium) will then according to the protocol have a transesophageal echocardiogram (TEE) to show the eventual mechanism of the shunt. If the TEE will not show any signs of a residual shunt, the patients will undergo a computed tomography angiogram (CTA) of the pulmonary circulation to exclude arterio-venous fistulas as a cause of the shunt seen on TTE. The investigators will also show the comparison in functional closure between classic and alternative device occluders.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a neurological event confirmed by a neurologist.
* Patients who underwent percutaneous closure of PFO in MC Medicor (Slovenia) from 2006 to 2022.

Exclusion Criteria:

* Patients who had additional congenital heart defects (as is atrial septal defects).
* Professional divers, who had the percutaneous closure of PFO because of an episode of decompression sickness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included patients who met our inclusion criteria, regardless of age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-07-11 (Estimated); Study Completion 2024-07-11 (Estimated)

PRIMARY OUTCOMES:
CVI | From date of percutaneous closure until the date of the last contrast transthoracic echocardiogram, assessed up to 24 months.
  Cerebrovascular insult
TIA | From date of percutaneous closure until the date of the last contrast transthoracic echocardiogram, assessed up to 24 months.
  Transient ischemic attack
Death | From date of percutaneous closure until the date of death from any cause.
  From cardiac and non-cardiac reasons

SECONDARY OUTCOMES:
AF | From date of percutaneous closure until the date of the last contrast transthoracic echocardiogram, assessed up to 24 months.
  Atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Marjeta Zorc, MD, PhD, Study Chair — MC Medicor; Marko Noc, MD, PhD, Study Director — MC Medicor
Locations (1):
- MC Medicor, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: During the period of 24 months.
Access Criteria: The Clinical Trials ID of the study.